CLINICAL TRIAL: NCT03895060
Title: Vertical and Horizontal Alveolar Ridge Augmentation Using Autogenous Onlay Ring Blocks Combined With Simultaneous Guided Bone Regeneration Using Native Collagen Membrane in Atrophic Anterior Maxilla.
Brief Title: Vertical and Horizontal Alveolar Ridge Augmentation Using Autogenous Onlay Blocks Combined With Guided Bone Regeneration Using Native Collagen Membrane in Atrophic Anterior Maxilla.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Moemen Abdel Salam Dewedar, Principal Investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOI CairoU
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Anterior Maxilla With Deficient Ridge Height and/or Width

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- autogenous ring blockls with GBR covered by collagen membrane (Experimental): Vertical and horizontal ridge augmentation using autogenous onlay ring blocks combined with simultaneous guided bone regeneration using native collagen membrane in atrophic anterior maxilla.
  Interventions: Device: autogenous ring blockls with GBR covered by collagen membrane

INTERVENTIONS:
Device: autogenous ring blockls with GBR covered by collagen membrane — * A crestal incision is made using No. 15 blade extending over the anterior maxilla, an anterior vertical releasing incision is made and a full mucoperiosteum flaps elevated to provide access to the alveolar ridge and the lateral aspect of the maxilla
  * Autogenous onlay ring blocks is taken by a trephine bur from the chin area and then fixed by screws to the deficient maxillary alveolar height.
  * Equally autogenous and xenograft bone particles is packed around the screw to fill the defect area completely.
  * The collagen membrane is fixed to the alveolar ridge by bone tacks and the mixture of autogenous and xenograft bone is then packed.
  * The flap will then be closed using interrupted 4/0 resorbable sutures.

SUMMARY:
Many different techniques exist for effective vertical bone augmentation, such as the use of particulate bone grafts and bone graft substitutes, barrier membranes for guided bone regeneration (GBR), autogenous and allogenic block grafts, and the application of distraction osteogenesis. Harvesting of autogenous block grafts is associated with greater morbidity compared with the less invasive procedure of using autogenous particles harvested through bone scrapers. On the other hand, particulate grafts always require a space-maintaining barrier, or their physical properties would not allow three-dimensional bone regeneration as those of block grafts do.

DETAILED DESCRIPTION:
An autogenous ring block is harvested from the chin area by trephine bur and the autogenous bone chips will be collected with a bone scraper, then a specially manufactured machine titanium tenting screw is used to fasten the ring block to the alveolar ridge. Two or three ring blocks is screwed according to the defect. Then resorbable collagen membrane is fixed to the alveolar ridge instead of the titanium-reinforced e-PTFE and equally autogenous and xenograft bone particles is packed around the screw to fill the defect area completely. Extreme care is taken to avoid autogenous particles drifting distally toward the area of the block. The barrier membrane was then closed over the block and particulate graft and fixed by bone tacks. Then periosteal releasing incision is done to allow tension free adaption of the mucoperisteal flap.

ELIGIBILITY:
Inclusion Criteria:

* Patients with partially edentulous in the anterior area of the maxilla, with a residual ridge that allowed insertion of ≤11.5 mm length implants.
* Both sexes.
* No intraoral soft and hard tissue pathology
* No systemic condition that contraindicate implant placement.

Exclusion Criteria:

* Pathology.
* Heavy smokers more than 20 cigarettes per day.
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems
* Disorders to implant are related to history of radiation therapy to the head and neck neoplasia, or bone augmentation to implant site
* Immunodeficiency pathology, bruxism, stress situation (socially or professionally), emotional instability, and unrealistic aesthetic demands.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Bone gained vertically | 6 months
  Amount of bone gained vertically will be measured using CBCT